CLINICAL TRIAL: NCT06552819
Title: User Experience of a Gait Training Treadmill for Home Rehabilitation of Children With Chronic Conditions
Acronym: EMMVIES-UX
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC24_0261
Record Dates: First submitted 2024-08-06; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Chronic Diseases in Children
Keywords: User experience, home program, treadmill, virtual reality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cerebral palsy, obesity and neuromuscular disease, parents and therapists
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
"In the context of limited accessibility to prolonged and efficient rehabilitation programs based on physical activity, this study aims to develop a home program for children with chronic diseases affecting physical health (including cerebral palsy, obesity, and neuromuscular diseases). The French company EzyGain has designed a compact treadmill equipped with sensors and a safety system, which communicates with a tablet application and a virtual reality headset to support at-home rehabilitation. This study seeks to advance the development of this solution into a prolonged and progressive training program, tailored to positively impact children's health. Future users, including children, their parents, and therapists, will be at the heart of the development process. A qualitative methodology will be employed, incorporating focus groups and a series of user experience (UX) questionnaires. The research hypothesis is that user feedbacks will enable the development of an appropriate solution that meets their specific needs and ensures high adoption rates of the device.

This study is the first step before assessing the impact of the solution in these 3 groups of children (with cerebral palsy, obesity and neuromuscular disease)."

DETAILED DESCRIPTION:
"Visit 1: Children, accompanied by one of their parents, will test the treadmill and the associated rehabilitation games on a tablet and in immersive virtual reality in its current version, and UX questionnaires will be administered.

Visit 2: Children, parents, and therapists, in groups of 6 to 8, will participate in focus groups during which they will express their opinions regarding the solution they tested in Visit 1 and discuss areas for improvement.

(several monthsare dedicated to the developpement of the solution by the society, based on the children, parents and therapists' feedbacks)

Visit 3: Children, accompanied by one of their parents, will test the treadmill and the associated rehabilitation games on a tablet and in immersive virtual reality in its new version, and UX questionnaires will be administered."

ELIGIBILITY:
"Inclusion Criteria for the children:

* aged between 8 and 18 years old
* capable of walking during 5 minutes on a treadmill with or without walking aid, and with or without body weight support
* diagnosis of one the following pathology: bilateral cerebral palsy, obesity, spinal muscular amiotrophy type 3, Duchenne, congenital myopathy, Charcot Marie Tooth
* Gross Motor Function Classification System (GMFCS) I to III for the children with cerebral palsy
* IMC superior to the centile IOTF-30 for the children with obesity
* Functionnal level of 2 to 6 on the Walton scale, or 3 to 7 on the Vignos scale for the children with neuromuscular disease

Inclusion Criteria for the parents:

- parent of an eligible child

Inclusion Criteria for the therapists:

- Therapist of at least one eligible child

Inclusion Criteria for all:

* Able to express oneself and respond to a questionnaire in French
* Formulate their non-opposition to participate in the research

Exclusion Criteria:

* Deprived of liberty by judicial or administrative decision
* Subject to a legal protection measure"

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients and parents from the active lists of medical doctors of the structures involved in the project. Therapists of the structures involved in the project.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Focus group outputs | Between the second and third week
  List of topics addressed during the focus groups by patients, parents, and therapists. The topics will include: the needs and expectations of an at-home rehabilitation tool including virtual reality, perceived barriers and facilitators, and acceptability related to certain features of the solution.

SECONDARY OUTCOMES:
User Experience Questionnaire (UEQ-S) | Day 1 and 6 months
  UX will be evaluated using the French short version of the User Experience Questionnaire (UEQ-S). It contains 8 items grouped into two scales: pragmatic qualities (efficiency, clarity, dependability) and hedonic qualities (stimulation, novelty). The format of the items is a semantic differential (e.g., Complicated - Simple) with a 7-point Likert scale.
Usability Metric for User Experience (UMUX) | Day 1 and 6 months
  Usability will be evaluated using the French version of the Usability Metric for User Experience (UMUX). The UMUX is a short 4-item questionnaire. The items are statements regarding ease of use and usefulness, with which respondents express their agreement on a 7-point Likert scale. Scores obtained from the UMUX will allow positioning the usability of the solution on the SUS interpretation scale (""worst imaginable"", ""poor"", ""acceptable"", ""good"", ""excellent"", or ""best imaginable"").
Ease with technology | Day 1 and 6 months
  Ease with technology will be assessed by the following question: ""On a scale of 1 to 10, how do you rate your ease with technologies?""
Cybersickness | Day 1 and 6 months
  Cybersickness will be evaluated using the Virtual Reality Sickness Questionnaire (VRSQ) which measures motion sickness-like sensations resulting from the use of virtual reality headsets. Participants rate the severity of each of the 9 VRSQ items from 0 to 3 (none, mild, moderate, severe). The total score reflects the average of the oculomotor discomfort and disorientation scores on a scale of 100. An internal questionnaire covering aspects of comfort, enjoyment, presence in the virtual environment (VE), and immersion will be used to inquire about participants' experiences with the VE and the VR headset. Participants respond on a visual analog scale from 0 to 10.
Children's perception of the games | Day 1 and 6 months
  Children's perception of the games will be assessed using an internal questionnaire inspired by the Game User Experience Satisfaction Scale (GUESS). The items are statements with which respondents express their agreement on a 7-point Likert scale. The scores for the various items will be summed and will allow the company to identify the most appreciated games and the weaknesses of others.
Acceptability | Day 1 and 6 months
  The acceptability from the perspective of the therapist or parent will be assessed using an internal questionnaire . The questions include their evaluations of the child's movement behavior, the level of support needed, engagement during the session, and their opinion on the use of virtual reality on a 5-point Likert scale."

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, Maine Et Loire, France

IPD SHARING:
Plan to Share IPD: No